CLINICAL TRIAL: NCT03554811
Title: Early Rehabilitation Using Functional Electrical Stimulation Assisted Supine Cycling Effect on Muscle Mass, Strength, Biomarkers, and Functional Outcomes as Compared With Conventional Exercise and Early Mobilization Alone in Critically Ill Patients in the Intensive Care Unit
Brief Title: Early Rehabilitation Using Functional Electrical Stimulation Assisted Supine Cycling in the Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fresno Community Hospital and Medical Center (Other)
Collaborators: Western University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018015
Record Dates: First submitted 2018-05-20; First posted 2018-06-13 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: ICU Acquired Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Functional electrical stimulation assisted supine cycling (Experimental): Patients will start functional electrical stimulation assisted supine cycling (FESC) within 48 hours of ICU admission and will undergo up to 1 hour of supine cycling daily, 5 days per week for 28 days, or until discharge from ICU.
  Interventions: Device: Functional electrical stimulation assisted supine cycling (FESC); Other: Conventional early exercise and mobility interventions
- Conventional early exercise and mobility interventions (Active Comparator): Patients will undergo standard ICU exercise and mobility interventions.
  Interventions: Other: Conventional early exercise and mobility interventions

INTERVENTIONS:
Device: Functional electrical stimulation assisted supine cycling (FESC) — A supine cycle ergometer attached to a six-channel stimulator will be used for FESC. Surface electrodes will be applied to the hamstrings, quadriceps, and calf muscles on both legs. Muscles will be stimulated at specific stages throughout the cycling phase. Each session will start with a 1 minute motor-driven passive cycling warm-up at a rate of 20 revolutions per minute. Patients will continue with passive, active-assisted, or active cycling, according to their level of participation. If the patients stop cycling actively, the ergometer will revert to passive cycling.
  Arms: Functional electrical stimulation assisted supine cycling
Other: Conventional early exercise and mobility interventions — These interventions will be based on the patient's alertness and medical stability, and includes activities to maintain or increase limb range of motion and strength, in and out of bed mobility, sit to stand, and transfer training, as well as assisted ambulation.

SUMMARY:
Critically ill patients in the intensive care unit are known to lose muscle mass and function at a rapid rate. Currently, there is a global recognition and shift in the ICU culture to reduce sedation and encourage exercise and mobilization early during the ICU stay. Functional stimulation assisted supine cycling can be applied to patients in the bed and does not require patient participation. This study seeks to evaluate the effect of conventional exercise and early mobilization in combination with functional stimulation assisted supine cycling applied early during the ICU on muscle mass, strength, and physical function, as well as patient-reported disability as compared to conventional exercise and early mobilization alone.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Admitted to the ICU with a predicted ICU length of stay ≥ 4 days
* Expected to survive the ICU stay
* Expected to receive mechanical ventilation > 48 hours
* Able to perform physical outcome measures pre-morbidly (with or without an assisted device)

Exclusion Criteria:

* Proven or suspected neuromuscular weakness affecting the legs (eg- stroke or Guillain-Barré syndrome)
* Lower limb amputation(s)
* Assessed by medical staff as approaching imminent death or withdrawal of medical treatment within 36 hours
* Pregnancy
* Body mass index > 40
* Presence of external fixator or superficial metal in lower limb
* Open wounds or skin abrasions at electrode application points
* Presence of pacemaker or implanted defibrillator
* Transferred from another ICU after >48 hours of consecutive mechanical ventilation
* Lower limb malignancy
* Pre-existing intellectual disability or cognitive impairment limiting the ability to accurately follow instructions
* Body habitus unable to fit the bike
* Palliative goals of care
* Unable to participate in FESC within 48 hours of ICU admission due to logistic reasons or due to failure in daily screening for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change of rectus femoris cross-sectional area | Baseline (within 24 hours of enrollment), weekly during ICU admission (up to a maximum of 28 days), at ICU discharge (an average of 11 days after admission), and at hospital discharge (an average of 15 days after admission)
  Ultrasound measurements will be done with patients in supine position with their leg in passive extension and neutral rotation.

SECONDARY OUTCOMES:
Diaphragm muscle thickness | Baseline (within 24 hours of enrollment), weekly in the ICU (up to a maximum of 28 days), at ICU discharge (an average of 11 days after admission), and at hospital discharge (an average of 15 days after admission)
  Thickness will be measured by ultrasound at the zone of apposition during inspiration or expiration using the intercostal approach.
Muscle strength | Baseline (within 24 hours of enrollment), weekly in the ICU (up to a maximum of 28 days), at ICU and hospital discharge (an average of 11 and 15 days after admission, respectively), and at 90 days, 6 months, and 1 year post ICU discharge
  Muscle strength will be assessed using the Medical Research Council Scale. This muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle. Weaker muscles will range from 0-3 and stronger muscles will receive grades 4 or 5.
Muscle strength | Baseline (within 24 hours of enrollment), weekly in the ICU (up to a maximum of 28 days), at ICU and hospital discharge (an average of 11 and 15 days after admission, respectively), and at 90 days, 6 months, and 1 year post ICU discharge
  Muscle strength will be assessed using hand-held dynamometry
Physical function | Baseline (within 24 hours of enrollment), weekly during ICU admission (up to a maximum of 28 days), at ICU discharge (an average of 11 days after admission), and at hospital discharge (an average of 15 days after admission)
  Physical function will be assessed using the physical function in ICU (PFIT) test
Physical function | Baseline (within 24 hours of enrollment), weekly during ICU admission (up to a maximum of 28 days), at ICU discharge (an average of 11 days after admission), and at hospital discharge (an average of 15 days after admission)
  Physical function will be assessed using the functional status score in the ICU (FSS-ICU). This score consists of 3 pre-ambulation categories (rolling; supine to sit transfer; and unsupported sitting) and 2 ambulation categories (sit to stand transfers; ambulation). Each category is scored from 1 (total dependent assistance) to 7 (complete independence) with a total score range of 0-35 (0: unable to perform a task due to physical limitations or medical status).
Physical function | Baseline (within 24 hours of enrollment), weekly during ICU admission (up to a maximum of 28 days), at ICU discharge (an average of 11 days after admission), and at hospital discharge (an average of 15 days after admission)
  Physical function will be assessed using the short physical performance battery (SPPB)
Physical function | Baseline (within 24 hours of enrollment), weekly during ICU admission (up to a maximum of 28 days), at ICU discharge (an average of 11 days after admission), and at hospital discharge (an average of 15 days after admission)
  Physical function will be assessed using the six-minute walk test (6MWT)
Quality of life | At hospital discharge (an average of 15 days after admission), and 90 days, 6 months, and 1 year post ICU discharge
  Quality of life will be measured using the 36-item Short Health Survey (SF-36), which assess eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a 0-100 scale and items in the same category are averaged together to create the 8 scale scores, with 0 being the lowest score and 100 being the highest for each category.
Cognition | At hospital discharge (an average of 15 days after admission)
  Cognition will be assessed using the Montreal Cognitive Assessment (MoCA).
Hospital length of stay | Through hospital discharge, an average of 15 days
  The total hospital length of stay for this admission will be calculated.
ICU length of stay | Through ICU discharge, an average of 11 days
  The total ICU length of stay for this admission will be calculated.
Duration of mechanical ventilation | Through discontinuation of mechanical ventilation, an average of 10 days
  The total length of time on mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Smith, PT, DPT, Principal Investigator — Community Medical Centers
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No